CLINICAL TRIAL: NCT05309811
Title: Effect of Repeated Low-Level Red-Light Therapy on Visual Field Damage in Primary Open-angle Glaucoma: A Randomized Cross-over Clinical Trial
Brief Title: Effect of Repeated Low-Level Red-Light Therapy on Visual Field Damage in Primary Open-angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020KYPJ108
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Open Angle Glaucoma; Eye Diseases
Keywords: Open-angle glaucoma; Repeated low-level red-light therapy; Visual field
MeSH Terms: conditions — Glaucoma, Open-Angle; Eye Diseases | interventions — Antiglaucoma Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): RLRL therapy with routine IOP-lowering medications in the 1st-12th weeks then crossing to only routine IOP-lowering medications in the 13th-24th weeks
  Interventions: Device: RLRL therapy; Drug: Routine IOP-lowering medications
- Group B (Experimental): Only routine IOP-lowering medications in the 1st-12th weeks then crossing to RLRL therapy with routine IOP-lowering medications in the 13th-24th weeks
  Interventions: Device: RLRL therapy; Drug: Routine IOP-lowering medications

INTERVENTIONS:
Device: RLRL therapy — Each RLRL treatment lasts three minutes. RLRL treatments will be performed twice a day, with at least four hours between each RLRL treatment.
  Other Names: Repeated Low-Level Red-Light Therapy
Drug: Routine IOP-lowering medications — Medications prescribed for IOP control by glaucoma specialists in the outpatient.
  Other Names: Anti-glaucoma medications

SUMMARY:
The purpose of this study is to investigate the effect of repeated low-level red-light therapy on existing visual field damages in primary open-angle glaucoma patients.

DETAILED DESCRIPTION:
Glaucoma is one of the main causes of visual impairment worldwide. Elevated intraocular pressure (IOP) is an important risk factor for glaucoma and the majority of anti-glaucoma therapies focus on the control of IOP. However, IOP-lowering treatments cannot directly attenuate optic neurodegeneration and rescue vulnerable retinal ganglion cells (RGCs). The glaucomatous symptoms could continue to deteriorate in some patients after optimal IOP control, which highlighted the need for alternative therapies targeting neuroprotection.

Chronic ischemia is another potential factor in the pathogenesis of glaucoma. Clinical trials suggested that calcium channel blockers such as nilvadipine could increase ocular blood flow and postpone visual field deterioration in normal-tension glaucoma. Furthermore, it was found that Ginkgo biloba extract, another vasoactive drug, could reverse existing visual field damages, which indicated that improved ocular circulation would salvage dysfunctional RGCs and its efficacy could be observed in a relatively short time frame.

The repeated low-level red-light (RLRL) therapy has regulatory effects on blood supply, which provides an innovative and non-invasive approach for the treatment of glaucoma. Considering the possible ischemic mechanism of POAG, it is expected that RLRL therapy could improve ocular circulation and reverse compromised visual functions. Using a randomized clinical trial with cross-over design, the purpose of this study is to investigate the effect of RLRL therapy on existing visual field damages in POAG patients.

This study is a 24-week, prospective, randomized, cross-over clinical trial, enrolling POAG patients with well-controlled IOP as participants. Study participants will be randomly allocated to two groups, with one group receiving RLRL therapy from the 1st to the 12th week and the other receiving RLRL therapy from the 13th to the 24th week. Use of IOP-lowering medications is allowed throughout the 24 weeks. An interim analysis to ensure the safety of RLRL therapy is scheduled after the 12th week. Linear mixed models will be used to determine changes in visual field and assess other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-69 years;
2. Diagnosis of primary open-angle glaucoma with definite visual field defects in either eye (MD <-3dB);
3. Well-controlled IOP in both eyes (IOP<21mmHg).

Exclusion Criteria:

1. Severe visual field defects in either eye (MD <-22dB);
2. Visual field defects caused by other diseases in either eye;
3. Unreliable results of visual field or IOP measurements in either eye;
4. Diagnosis of other ocular diseases in active phase in either eye;
5. History of refractive surgeries in either eye;
6. History of other ophthalmic laser treatments or intraocular surgeries in the last 3 months in either eye;
7. Refusing to inform consents or having difficulties to take part in follow-ups in next 6 months.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes of mean deviations (MD) in visual field tests | 12 weeks and 24 weeks
  The twelve-week changes of MD are characterized as differences between the 12-week follow-up visit and the baseline visit or differences between the 24-week visit and the 12-week follow-up visit. The Humphrey Visual Field Analyzer will be used to measure MD (dB).

SECONDARY OUTCOMES:
Changes of mean deviations (MD) in visual field tests | 4 weeks and 16 weeks
  The four-week changes of MD are characterized as differences between the 4-week follow-up visit and the baseline visit or differences between the 16-week visit and the 12-week follow-up visit.
  The Humphrey Visual Field Analyzer will be used to measure MD (dB).
Incidence rates of significant reversal of visual field damages | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week incidence rates of significant reversal of visual field damages are rates of POAG patients with MD reversal ≥ 3dB between the 4-/12week follow-up visits and the baseline visit or between the 16-/24-week follow-up visits and the 12-week follow-up visit.
  The Humphrey Visual Field Analyzer will be used to measure MD (dB).
Changes of pattern standard deviations (PSD) in visual field tests | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week changes of PSD are characterized as differences between the 4-/12week follow-up visit and the baseline visit or differences between the 16-/24-week visit and the 12-week follow-up visit.
  The Humphrey Visual Field Analyzer will be used to measure PSD (dB).
Changes of the thickness of parapapillary retinal nerve fiber layer | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week changes of the thickness of parapapillary retinal nerve fiber layer (RNFL) are characterized as differences between the 4-/12week follow-up visits and the baseline visit or differences between the 16-/24-week follow-up visits and the 12-week follow-up visit.
  Spectralis HRA OCT and Optovue OCT will be used to measure the thickness of parapapillary RNFL (μm).
Changes of the thickness of perifoveal ganglion cell-inner plexiform layer | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week changes of the thickness of perifoveal ganglion cell-inner plexiform (CG-IPL) are characterized as differences between the 4-/12week follow-up visits and the baseline visit or differences between the 16-/24-week follow-up visits and the 12-week follow-up visit.
  Spectralis HRA OCT and Optovue OCT will be used to measure the thickness of perifoveal CG-IPL (μm).
Changes of the thickness of central macular choroid | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week changes of the thickness of central macular choroid are characterized as differences between the 4-/12week follow-up visits and the baseline visit or differences between the 16-/24-week follow-up visits and the 12-week follow-up visit.
  DRI OCT Triton and Optovue OCT will will be used to measure the thickness of central macular choroid (μm).
Changes of the parapapillary capillary density | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week changes of parapapillary capillary density (CD) are characterized as differences between the 4-/12week follow-up visits and the baseline visit or differences between the 16-/24-week follow-up visits and the 12-week follow-up visit.
  DRI OCT Triton and Optovue OCT will will be used to measure parapapillary CD (%).
Change of the perifoveal capillary density | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week changes of perifoveal capillary density (CD) are characterized as differences between the 4-/12week follow-up visits and the baseline visit or differences between the 16-/24-week follow-up visits and the 12-week follow-up visit.
  DRI OCT Triton and Optovue OCT will be used to measure perifoveal CD (%).
Incidence rates of treatment-emergent adverse events | 4 weeks, 12 weeks, 16 weeks and 24 weeks
  The four-week and twelve-week incidence rates of treatment-emergent adverse events are rates of treatment-emergent adverse events between the 4-/12week follow-up visits and the baseline visit or between the 16-/24-week follow-up visits and the 12-week follow-up visit. Subjects will be asked to report any treatment-emergent adverse event, including but not limited to glare, flash blindness, and afterimages.

CONTACTS AND LOCATIONS:
Overall Officials: Mingguang He, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes